CLINICAL TRIAL: NCT05726643
Title: Effect of Kinesiotaping Augmented By Resistive Exercise on Fatigue, Physical Strength, Quality of Life in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mos'ad Ebrahim Rmdan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alaa_Negm_MSc_2023
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Fatigue; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistive training group (Active Comparator): consists of 20 patients who will receive resistive training for 2times per week for 12 weeks
  Interventions: Other: resistive training
- kinesotaping group (Experimental): consists of 20 patients who will receive resistive training program augmented by kinesotaping, 2 times /week for 12 weeks.
  Interventions: Other: resistive training; Other: kinesiotaping

INTERVENTIONS:
Other: resistive training — 5 minutes warming up exercise for various parts of the body as moderately energetic walking.
  5 to 10 minutes stretching exercise for (pectorals major, hamstring, hip flexors, and calf muscles) with each static stretch held for at least 20 seconds in first week and then 30 seconds for the remaining 5 weeks and this will be repeated about four times.
  10 to 15 minutes strengthening exercise by using weights for lower limbs (knee extensors, hip abductors, and hip extensors) at first session for each patient. Ten repetitions maximum (10 RM) will be determined, which is the maximal weight can be lifted through the entire range of motion 10 times.
Other: kinesiotaping — Tape will be applied to each participant in the treatment group for the sartorius, rectus femoris, hamstrings, tibialis anterior, fibularis brevis, and the patella bilaterally using strips of the standard 2-inch Kinesio Tex Tape. The first and last inch of each strip will be applied without tension. The length of the strip will be applied with a 20%- 25% stretch and downward pressure to the insertion. Each of the sartorius, rectus femoris, hamstrings, tibialis anterior and fibularis brevis tapings used an I-strip. AY strip will be utilized for the patellar taping.
  Arms: kinesotaping group

SUMMARY:
The purpose of the study will be to investigate the effect of kinesotaping augmented by resistive exercise on fatigue, muscle strength, and QoL in breast cancer survivors.

DETAILED DESCRIPTION:
The present study will provide an evidence base to women's health care providers about the effect of strength training augmented by kinesotaping on fatigue, QoL and muscle strength in breast cancer women compared to strength training alone

ELIGIBILITY:
Inclusion Criteria:

* Patient's age will range from 40- 55 years.
* Their body mass index (BMI) will be from 25 to 29,9 Kg/m2.
* They suffer from breast cancer.
* They will receive chemotherapy within previous 3 months.
* They complain from fatigue, deterioration in their daily living activity (ADL) and feeling of weakness in their muscles.

Exclusion Criteria:

* Respiratory or heart problems affecting mobility
* Marked skeletal deformity.
* Visual system affection.
* Cognition problems.
* Previous surgeries at their back and/or lower limbs.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in fatigue | at baseline and after 12 weeks of intervention
  The Fatigue Severity Scale is a 14-item will be used to measure the severity, frequency and diurnal variation of fatigue, as well as its perceived interference with quality of life.
Assessing the change in quality of life | at baseline and after 12 weeks of intervention
  By using 36-Item Short Form (SF-36) health survey will be used to assess QoL. The SF-36 questionnaire includes eight multiple-item subscales that evaluate physical function, social functioning, role limitations due to physical problems and role limitations due to emotional problems, mental health, vitality, pain and general health perception. Total score on each SF-36 subscale ranges between 0 and 100. Greater score indicates better QoL
Assessing the change in muscle strength | at baseline and after 12 weeks of intervention
  Muscle strength will be assessed using dynamometer at starting and after 12 weeks of the treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Negm, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physica therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided